CLINICAL TRIAL: NCT02332187
Title: Effect of All-Stim 2 Quadriceps Treatments on Limb Muscle Strength In Mechanically Ventilated Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer have resources to complete this work.
Sponsor: Gerald Supinski (Other)
Responsible Party: Sponsor-Investigator, Gerald Supinski, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 12-0807-F6A
Record Dates: First submitted 2014-12-30; First posted 2015-01-06 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Weakness
MeSH Terms: conditions — Asthenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham electrical stimulation (Sham Comparator): The intervention will consist of sham electrical stimulation using an All Stim stimulator of each quadriceps leg muscle for 30 minutes per day for a total of 7 days.
  Interventions: Device: Sham electrical stimulation using an All Stim stimulator
- Active electrical stimulation (Active Comparator): The intervention will consist of active electrical stimulation using an All Stim stimulator of each quadriceps leg muscle for 30 minutes per day for a total of 7 days.
  Interventions: Device: Active electrical stimulation using an All Stim stimulator

INTERVENTIONS:
Device: Active electrical stimulation using an All Stim stimulator — This is an FDA approved stimulator that is used for strengthening the quadriceps muscle.
  Arms: Active electrical stimulation
Device: Sham electrical stimulation using an All Stim stimulator — With this intervention the All Stim unit is turned off and no electrical stimulation is provided.
  Arms: Sham electrical stimulation

SUMMARY:
Patients that are on mechanical ventilators in medical intensive care units (MICU) have extremely weak leg muscles. Currently there is no treatment to prevent or reverse this weakness. Treatments with a thigh muscle stimulator, called an All Stim 2, can improve leg muscle strength and help patients regain leg function after knee surgery. The purpose of the present study is to determine if treatments with the All Stim 2 device can also improve leg muscle strength in patients on mechanical ventilation.

DETAILED DESCRIPTION:
The objective for this study is to determine if daily exercise using All-Stim 2 stimulation of quadriceps muscles will increase leg strength and improve outcomes (duration of hospitalization, long term mobility, long term disability) for mechanically ventilated MICU patients. The investigators plan to randomize patients accepted into this protocol to administration of either sham exercise (i.e. placement of All-Stim 2 units on the legs for 30 minutes a day without activation of the electrical stimulation program) or active exercise (placement of All-Stim 2 electrodes on both legs and stimulating quadriceps muscles to rhythmically contract for 30 minutes a day). The two groups (sham and active exercise) will be treated for 30 minutes a day for seven days. The effects of exercise on quadriceps strength will be assessed by measuring quadriceps force generation (QuadTw) in response to magnetic stimulation of the femoral nerves. The QuadTw assessment will be made immediately before institution of sham or active exercise and will repeated one day after the conclusion of the seven day training regimen. Chart review and patient follow-up will be used to determine if this treatment regimen also has an impact on clinical outcome measures, i.e. duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring mechanical ventilation for more than 48 hours
* Respiratory failure present

Exclusion Criteria:

* The physician caring for the patient determines that the patient is too unstable
* Use of high dose pressors (more than 15 mcg/min of norepinephrine or more than 15 mg/kg/min of dopamine)
* Use of more than 80% FiO2 (fractional concentration of oxygen) or more than 15 cm H2O (water) of PEEP (positive end expiratory pressure)
* Presence of a cardiac pacemaker or implanted defibrillator
* Use of neuromuscular blocking agents within the 48 hours preceding testing
* History of a preexisting neuromuscular disease
* Presence of profound and uncorrectable hypokalemia (less than 2.5) or hypophosphatemia (less than 1.0)
* Pregnancy
* If the patient is a prisoner
* If the patient is institutionalized
* If it is thought that the patient will have care withdrawn within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S Supinski, MD, Principal Investigator — University of Kentucky
Locations (1):
- Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified data to other researchers on request. We cannot, however, under the terms of our IRB approval, provide primary data which contains information that may identify participants. Data will be released once the paper is accepted for publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2019
Access Criteria: Any researcher associated with a University or Pharmaceutical company

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Electrical Stimulation | Active Electrical Stimulation
Started | 5 | 10
Completed | 3 | 7
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Electrical Stimulation | Active Electrical Stimulation | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (15.5) | 46.1 (15.5) | 50.2 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 10 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Quadriceps Muscle Strength
Description: The investigators will measure quadriceps leg strength before and after one week of either sham or active electrical stimulation of the quadriceps muscle.
Time Frame: Baseline and One week
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Sham Electrical Stimulation | Active Electrical Stimulation
Number analyzed (Participants) | 3 | 7
Newtons
  Right quadricep | -5.0 (5.8) | 2.6 (2.2)
  Left quadricep | -6.1 (7.4) | 3.4 (3.6)

2. Secondary Outcome: Duration of Hospitilization
Description: The investigators will record the total time patients remain hospitilized after entry into the study.
Time Frame: Baseline to discharge in weeks, up to five weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Sham Electrical Stimulation | Active Electrical Stimulation
Number analyzed (Participants) | 3 | 7
weeks | 4.6 (0) | 3.0 (0.7)

ADVERSE EVENTS:
Time Frame: Baseline to end of hospitalizations for all participants, up to five weeks.
Arm/Group | Sham Electrical Stimulation | Active Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Electrical Stimulation (N=5) | Active Electrical Stimulation (N=10)
Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT02332187/Prot_SAP_ICF_000.pdf